CLINICAL TRIAL: NCT06466447
Title: Effectiveness of Video Teletherapy in Treating Child and Adolescent Obsessive-Compulsive Disorder With Exposure and Response Prevention: a Retrospective Longitudinal Observational Study
Brief Title: Child and Adolescent OCD Outcomes From Exposure and Response Prevention Video Teletherapy Treatment
Status: Completed | Type: Observational
Sponsor: NOCD (Industry)
Responsible Party: Sponsor
Other Study IDs: NOCD002
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: exposure and response prevention; digital behavioral health; remote treatment; video therapy; children; adolescents
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obsessive-Compulsive Disorder: adolescents and children with obsessive-compulsive disorder
  Interventions: Behavioral: Exposure and response prevention therapy

INTERVENTIONS:
Behavioral: Exposure and response prevention therapy — Exposures and response prevention therapy (a type of cognitive-behavioral therapy for obsessive-compulsive disorder), delivered in real-time by therapists remotely via video. The treatment was augmented by between-session text messaging.

SUMMARY:
This is a naturalistic, observational study of children and adolescents with obsessive-compulsive disorder who were treated with exposure and response prevention via video teletherapy.

ELIGIBILITY:
Inclusion Criteria:

* obsessive-compulsive disorder

Exclusion Criteria:

* none

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a naturalistic sample of children and adolescents obsessive-compulsive disorder (OCD) who sought treatment for OCD from NOCD, Inc., a digital behavioral health company.
Sampling Method: Non-Probability Sample
Enrollment: 2173 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Dimensional Obsessive-Compulsive Scale | change from pre-treatment to post-treatment (after 11 weeks)
  self-rated psychometric instrument to measure symptom severity of multiple OCD subtypes (score range: 0-80)

SECONDARY OUTCOMES:
Depression Anxiety and Stress Scale (DASS-21) | pre-treatment, after 4 weeks, and post-treatment (after 11 weeks)
  self-rated psychometric instrument to measure depression, anxiety, and stress (score range: 0-63)

CONTACTS AND LOCATIONS:
Locations (1):
- NOCD, Inc., Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No